CLINICAL TRIAL: NCT02316236
Title: Effect of Dexmedetomidine on Outcomes During Emergence From Retroperitoneal Laparoscopic Surgery
Brief Title: Dexmedetomidine to Improve Outcomes During Emergence From Retroperitoneal Laparoscopic Surgery
Acronym: DEALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Dr, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-2014-6-22-01
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine loading dose (Experimental): dexmedetomidine is given at load dose
  Interventions: Drug: dexmedetomidine; Other: loading dose
- dexmedetomidine sustaining dose (Experimental): dexmedetomidine is given at sustaining dose
  Interventions: Drug: dexmedetomidine; Other: sustaining dose

INTERVENTIONS:
Drug: dexmedetomidine — an alpha-2 receptor agonist
  Other Names: dex
Other: loading dose — 0.8ug/kg of dexmedetomidine is given in 10 minutes
  Other Names: LD
  Arms: dexmedetomidine loading dose
Other: sustaining dose — 0.4ug/kg/min of dexmedetomidine is given
  Other Names: SD
  Arms: dexmedetomidine sustaining dose

SUMMARY:
The study is to observe whether dexmedetomidine could reduce agitation during emergence from general anesthesia in patients undergoing retroperitoneal laparoscopic surgery.

DETAILED DESCRIPTION:
Agitation during emergence is frequent after retroperitoneal urologic surgery. Dexmedetomidine is alpha-2 receptor agonist which shows sedative and algesic effect. In this study we will compare the effect of dexmedetomidine given by different protocols on emergence agitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for retroperitoneal laparoscopic surgery
* Patients with written informed consent

Exclusion Criteria:

* Patients with difficulty of communication
* Patients with risk of obstructive sleeping apnea syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2015-08-12 (Actual); Study Completion 2015-08-13 (Actual)

PRIMARY OUTCOMES:
Richmond Score | From end of sevoflurane inhalation to departure from PACU, an expected average of 1 hour

SECONDARY OUTCOMES:
Cough score | From end of sevoflurane inhalation to departure from PACU, an expected average of 1 hour
Time to awake | From end of sevoflurane inhalation to departure from PACU, an expected average of 1 hour
  time to open eyes to verbal command

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, PhD, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Yang S, Lee H. A dose-finding study of preoperative intravenous dexmedetomidine in children's emergence delirium after epiblepharon surgery. Eur J Ophthalmol. 2014 May-Jun;24(3):417-23. doi: 10.5301/ejo.5000396. Epub 2013 Nov 29. PMID 24338578
- [Result] Kim SY, Kim JM, Lee JH, Song BM, Koo BN. Efficacy of intraoperative dexmedetomidine infusion on emergence agitation and quality of recovery after nasal surgery. Br J Anaesth. 2013 Aug;111(2):222-8. doi: 10.1093/bja/aet056. Epub 2013 Mar 22. PMID 23524149
- [Result] Ibacache ME, Munoz HR, Brandes V, Morales AL. Single-dose dexmedetomidine reduces agitation after sevoflurane anesthesia in children. Anesth Analg. 2004 Jan;98(1):60-63. doi: 10.1213/01.ANE.0000094947.20838.8E. PMID 14693585